CLINICAL TRIAL: NCT04124640
Title: Observational Study in Real Life to Describe the Effectiveness of LIBICARE® in Women With Low Arousal and Sexual Desire Levels.
Brief Title: Observational Study in Real Life to Describe the Libicare® Effectiveness in Female Sexual Dysfunction.
Acronym: LIBIDOBS
Status: Completed | Type: Observational
Sponsor: Procare Health Iberia S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-LIB-2019-01
Record Dates: First submitted 2019-06-19; First posted 2019-10-11 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Female Sexual Dysfunction
MeSH Terms: interventions — Treatment Outcome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- treatment group: The study population will be women between 45 and 65 years old, both ages included, who present a decrease in sexual desire or arousal
  Interventions: Other: Patients' data (baseline characteristics, clinical and outcomes) from routine care visits

INTERVENTIONS:
Other: Patients' data (baseline characteristics, clinical and outcomes) from routine care visits — Use of a standardized scale to collect clinical and patient-centered data, to assess the effectiveness of Libicare in real life in female 45-65 years old. Patients' data (baseline characteristics, clinical and outcomes) will be collected according to sites routine care.

SUMMARY:
The decrease or absence sexual desire and arousal is the alteration of the sexual sphere that women most commonly refer to in adulthood and old age. Many women can refer a decrease or absence of desire and / or arousal without having the disorder typified in the DSM-5, but that can cause discomfort, worry and relationship problems in their day to day. Libicare® is a food supplement whose ingredients could have positive effects on the improvement of sexual function in women with low desire and arousal levels. The main ingredients of Libicare® are:

* Trigonella Foenum-graecum (Trigonella) (1)
* Tribulus Terrestris (Tribulus) (2)
* Turnera Diffusa (Damiana) (3)

DETAILED DESCRIPTION:
The main objective is to describe the effectivity of LIBICARE® in the improvement of desire and sexual arousal in women between 45 and 65 years old, in real life.

The secondary objectives of the study are:

* Evaluation of the 6 domains of the EVAS-M scale at 2 and 4 months of treatment.
* Assessment of the safety of LIBICARE® by collecting serious and non-serious adverse events.
* Evaluation of patient satisfaction with treatment at 2 and 4 months of treatment.
* Therapeutic compliance in taking the food supplement at 2 and 4 months of treatment.
* Study of the hormonal variation in relation to the values of total testosterone, free testosterone and SHBG, at the beginning, at 2 months and at 4 months of treatment, in those patients in which it is determined by routine clinical practice.
* To evaluate the degree of usefulness of the EVAS-M scale in clinical practice after 4 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women between 45 and 65 years old, both ages included.
* Women who refer decreased desire and / or sexual arousal.
* Women who will receive LIBICARE® by prescription of their doctor regardless of their participation or not in the study.
* Women who have given their informed consent in writing.

Exclusion Criteria:

* Women who suffer or have suffered breast cancer.
* Women in anticoagulant treatment.
* Women who, in the opinion of the researcher, cannot follow the study procedures.
* Women not be able to understand the nature of the study, the procedures to follow or who are not authorized to sign an informed consent
* Pregnant or lactating women
* Women with allergies to any of the components of Libicare®

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study population will be women between 45 and 65 years old, both ages included, who present a decrease in sexual desire or arousal
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
To describe the effectiveness of LIBICARE® in improving sexual desire and arousal in women between 45 and 65 years of age, in real life. | 4 month
  The effectiveness will be the increase in the score of the EVAS-M scale that will be provided to patients in the visita during the follow-up visits.

SECONDARY OUTCOMES:
Evaluation of the 6 domains of the EVAS-M scale at 2 and 4 months of treatment. | at 2 and 4 months of treatment
  Evaluation of the 6 domains of the EVAS-M scale ("Escala de Valoración de la Actividad Sexual en la mujer" in Spanish, score from 2 to 60 points) at 2 and 4 months of treatment
Evaluation of the safety of LIBICARE® by collecting serious and non-serious adverse events. | at 4 months of treatment
  The safety that will be defined by the serious and non-serious adverse reactions collected throughout the study.
Evaluation of patient satisfaction with treatment at 2 and 4 months of treatment. | at 2 and 4 months of treatment
  Evaluation of patient satisfaction with treatment using the Likert scale
Therapeutic compliance in taking the food supplement at 2 and 4 months of treatment. | at 2 and 4 months of treatment
  Therapeutic compliance will continue to be adjusted as much as possible to routine clinical practice using the Likert scale
Study of the hormonal variation in relation to the values of total testosterone, free testosterone and SHBG, at the beginning, at 2 months and at 4 months of treatment, in those patients in which it is determined by routine clinical practice. | at 0, 2 and 4 months of treatment
  Study of the hormonal variation in relation to the values of total testosterone, free testosterone and SHBG, at the beginning, at 2 months and at 4 months of treatment, in those patients in which it is determined by routine care
To evaluate the degree of usefulness of the EVAS-M (ESCALA DE VALORACION DE LA ACTIVIDAD SEXUAL in Spanish) scale in clinical practice after 4 months of treatment. | at 4 months
  Usefulness of using the EVAS-M scale in clinical practice (last visit)

CONTACTS AND LOCATIONS:
Overall Officials: Josep Combalia, MD, Study Director — Procare health Iberia; Santiago Palacios, Principal Investigator — Instituto Palacios de Salud y Medicina de la Mujer.
Locations (1):
- Instituto Palacios de Salud y Medicina de la Mujer, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rao A, Steels E, Beccaria G, Inder WJ, Vitetta L. Influence of a Specialized Trigonella foenum-graecum Seed Extract (Libifem), on Testosterone, Estradiol and Sexual Function in Healthy Menstruating Women, a Randomised Placebo Controlled Study. Phytother Res. 2015 Aug;29(8):1123-30. doi: 10.1002/ptr.5355. Epub 2015 Apr 24. PMID 25914334
- [Result] Akhtari E, Raisi F, Keshavarz M, Hosseini H, Sohrabvand F, Bioos S, Kamalinejad M, Ghobadi A. Tribulus terrestris for treatment of sexual dysfunction in women: randomized double-blind placebo - controlled study. Daru. 2014 Apr 28;22(1):40. doi: 10.1186/2008-2231-22-40. PMID 24773615
- [Result] Zhao J, Dasmahapatra AK, Khan SI, Khan IA. Anti-aromatase activity of the constituents from damiana (Turnera diffusa). J Ethnopharmacol. 2008 Dec 8;120(3):387-93. doi: 10.1016/j.jep.2008.09.016. Epub 2008 Sep 26. PMID 18948180